CLINICAL TRIAL: NCT03735719
Title: Biomarkers for Risk Stratification of Patients With ST-elevation Myocardial Infarction Treated With Primary Percutaneous Coronary Intervention
Brief Title: Biomarkers for Risk Stratification After STEMI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: BIOSTRAT
Record Dates: First submitted 2018-11-05; First posted 2018-11-08 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2018-11

CONDITIONS: Biomarkers; ST Segment Elevation Myocardial Infarction; Primary Percutaneous Coronary Intervention; Heart Diseases; Cardiovascular Diseases; Pathologic Processes; Heart Failure
Keywords: soluble ST2; galectin-3; prognosis; STEMI; primary PCI
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Heart Diseases; Cardiovascular Diseases; Pathologic Processes; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — From each patient will be collected 10 ml of venous blood which will be centrifugated to obtain serum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- STEMI patients: Patients with first STEMI treated with primary PCI are recruited in this study.
- Control group: The control group will consist of patients with risk factors for cardiovascular diseases, but without history of coronary artery disease or heart failure.

SUMMARY:
Despite modern reperfusion strategies, myocardial infarction leads to deleterious processes resulting in left ventricular remodelling (LVR) and heart failure (HF). Several biomarkers i.e. galectin-3 (Gal-3) and soluble ST-2 protein are involved in LVR as a result of inflammatory processes and fibrosis. There is an evidence of a high prognostic value of both biomarkers in prediction of outcomes in HF patients. This study will further investigate the role of Gal-3 and ST-2 in patients with ST-segment elevation myocardial infarction (STEMI) treated with primary percutaneous coronary intervention (PCI) and without prior HF in prediction of unfavourable outcomes.

DETAILED DESCRIPTION:
Heart failure is nowadays one of the leading problems in cardiology. Heart failure is associated with high morbidity and mortality, as well as high social costs, resulting mainly from a large number of hospitalizations. Galectin-3 and ST-2 have an important role in remodeling and fibrosis of the left ventricle, one of the key pathophysiological mechanisms leading to the development of heart failure. Galectin-3 is a protein secreted by activated macrophages, that stimulate inflammation and fibrosis of the myocardium. ST2 molecule is a soluble glycoprotein belonging to the family of interleukin-1 receptor, secreted by inflammatory cells, cardiomyocytes and endothelium. The ST2 has two clinically relevant isoforms - transmembrane (ST-2L, ST-2 ligand) and soluble (sST-2, soluble ST-2) circulating in the bloodstream. sST2 is present in the extracellular environment and through competitive binding with IL-33 prevents its connection with ST2L, and triggers myocardial fibrosis.

There is evidence of a prognostic value of both biomarkers in prediction of outcomes in heart failure patients. However, studies evaluating the role of Gal-3 and ST-2 in patients with ST-segment elevation myocardial infarction (STEMI) are lacking.

The study will include consecutive patients with first STEMI treated with percutaneous coronary intervention (PCI) in 1st Chair and Department of Cardiology, Medical University of Warsaw. The control group will consist of patients with risk factors for cardiovascular risk factors, but without history of coronary artery disease or heart failure. Patients will be followed for 12 months.

Blood will be sampled twice during the study: 72-96 hours after hospital admission and during a follow-up visit at 12 months. Blood will be collected for routine laboratory tests, Gal-3, ST-2 and other biomarkers: cardiac troponin I (cTnI), C-reactive protein (CRP) and N-terminal pro-B-type natriuretic peptide (NT-proBNP). Two-dimensional echocardiography will be performed 24-48 hours after PCI and during a follow-up visit at 12 months.

The aim of the study is to assess the prognostic value of Gal-3 and ST-2 in patients after first STEMI treated with PCI in prediction of left ventricular systolic and diastolic dysfunction, development of heart failure, need for cardiovascular hospitalization and death during one year follow-up after STEMI.

Furthermore, the baseline concentrations of biomarkers in the study and control groups will be compare.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years
* signed consent
* first STEMI treated with PCI

Exclusion Criteria:

* previous STEMI/non-STEMI,
* pre-existing HF,
* severe renal dysfunction (plasma creatinine level >220 mmol/L and/or creatinine clearance <30 mL/min),
* severe liver disease,
* chronic inflammatory disease,
* current neoplastic disease,
* life expectancy <1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study will include patients with first ST-elevation myocardial infarction treated with primary percutaneous coronary intervention.
Sampling Method: Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Biomarker-related risk stratification of heart failure occurrence after STEMI treated with PCI. | 12 months after STEMI
  Assessment of the prognostic value of Gal-3 and ST-2 in prediction of developing heart failure in one year observation after STEMI.
Biomarker-related risk stratification of one-year death occurrence after STEMI treated with PCI. | 12 months after STEMI
  Assessment of the prognostic value of Gal-3 and ST-2 in prediction of death in one year observation after STEMI.
Biomarker-related risk stratification of cardiovascular hospitalization occurrence after STEMI treated with PCI. | 12 months after STEMI
  Assessment of the prognostic value of Gal-3 and ST-2 in assessment of the risk of hospitalization for cardiovascular reasons in one year observation after STEMI.
Biomarker-related risk stratification of left ventricular systolic dysfunction occurrence after STEMI treated with PCI. | 12 months after STEMI
  Assessment of the prognostic value of Gal-3 and ST-2 in prediction of left ventricular systolic dysfunction in one year observation after STEMI.
Biomarker-related risk stratification of left ventricular diastolic dysfunction occurrence after STEMI treated with PCI. | 12 months after STEMI
  Assessment of the prognostic value of Gal-3 and ST-2 in prediction of left ventricular diastolic dysfunction in one year observation after STEMI.

SECONDARY OUTCOMES:
Correlation of serum biomarkers concentrations with cardiac remodeling | 12 months after STEMI
  Assessment of the correlation between Gal-3 and ST-2 with a size of an infarct scar and echocardiographic parameters
Correlation of serum biomarkers concentrations with a inflammation | 12-months observation
  Assessment of the correlation between Gal-3 and ST-2 with other biomarkers of inflammation (e.g C-reactive protein).
comparison to control subjects | baseline assessment
  Assessment of Gal-3 and ST-2 concentrations in comparison to the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Kapłon-Cieślicka, PhD, Study Chair — 1st Chair and Department of Cardiology, Medical University of Warsaw; Grzegorz Opolski, Professor, Study Chair — 1st Chair and Department of Cardiology, Medical University of Warsaw; Krzysztof J Filipiak, Professor, Study Chair — 1st Chair and Department of Cardiology, Medical University of Warsaw
Locations (1):
- 1st Chair and Department of Cardiology, Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided
The investigators will be able to share data for meta-analyses

REFERENCES:
- [Derived] Tyminska A, Kaplon-Cieslicka A, Ozieranski K, Budnik M, Wancerz A, Sypien P, Peller M, Balsam P, Opolski G, Filipiak KJ. Association of Galectin-3 and Soluble ST2, and Their Changes, with Echocardiographic Parameters and Development of Heart Failure after ST-Segment Elevation Myocardial Infarction. Dis Markers. 2019 Oct 10;2019:9529053. doi: 10.1155/2019/9529053. eCollection 2019. PMID 31687050
- [Derived] Tyminska A, Kaplon-Cieslicka A, Ozieranski K, Budnik M, Wancerz A, Sypien P, Peller M, Maksym J, Balsam P, Opolski G, Filipiak KJ. Association of galectin-3 and soluble ST2 with in-hospital and 1-year outcomes in patients with ST-segment elevation myocardial infarction treated with primary percutaneous coronary intervention. Pol Arch Intern Med. 2019 Nov 29;129(11):770-780. doi: 10.20452/pamw.15030. Epub 2019 Oct 23. PMID 31642446